CLINICAL TRIAL: NCT07407465
Title: Phase II Single Arm Study of Upfront Trastuzumab-Deruxtecan Plus Capecitabine and Bevacizumab for Patients With HER-2 Positive Metastatic Colorectal Cancer: the CHIMERA Study.
Brief Title: Upfront Trastuzumab-Deruxtecan Plus Capecitabine and Bevacizumab for Patients With HER-2 Positive Metastatic Colorectal Cancer.
Acronym: CHIMERA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIMERA; 2024-519479-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-10; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma; Rectal Adenocarcinoma; Rectal Cancer, Adenocarcinoma; Rectal Cancer, Metastatic; Colon Cancer Metastatic; Colon Cancer Adenocarcinoma
Keywords: colorectal cancer; HER-2 positive; Trastuzumab-deruxtecan; Capecitabine; Bevacizumab; mCRC
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms | interventions — trastuzumab deruxtecan; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trastuzumab-deruxtecan, capecitabine, bevacizumab (Experimental): * Trastuzumab-deruxtecan 5.4 mg/Kg, IV, d1 q3w;
  * Capecitabine 1000 mg/sqm B.I.D, oral, dd1-14 q3w;
  * Bevacizumab 7.5 mg/kg, IV, d1 q3w;
  Treatment will be received until progressive disease, unacceptable toxicity, consent withdrawal, investigator's decision or study termination, whichever occurs first.
  Interventions: Drug: Trastuzumab-Deruxtecan (T-DXd); Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Trastuzumab-Deruxtecan (T-DXd) — T-DXd at the dose of 5.4 mg/kg intravenous (as a 90 +/- 10 minute infusion) on day 1 every 3 weeks
Drug: Capecitabine — 1000 mg/sqm bis in die (BID) orally on days 1-14 every 3 weeks
Drug: Bevacizumab — 7.5 mg/kg intravenous (as a 30 minute infusion) on day 1 every 3 weeks

SUMMARY:
The aim of this study is to evaluate the activity of first-line trastuzumab-deruxtecan, capecitabine and bevacizumab in terms of overall response rate for patients with HER-2 positive metastatic/locally advanced unresectable colorectal cancer

DETAILED DESCRIPTION:
This is a multinational, Open-label, Single-arm Phase II trial in which patients with metastatic or locally advanced unresectable HER-2 positive colorectal cancer will receive upfront trastuzumab-deruxtecan, capecitabine and bevacizumab until progressive disease, unacceptable toxicity, consent withdrawal, investigator's decision or study termination, whichever occurs first. The primary endpoint of the study is Overall Response Rate by blinded independent central review. In order to preliminarily assess safety, a safety run-in phase will be conducted. The safety run-in phase will include the first 6 patients enrolled. After 6 patients will have received 3 cycles of study treatment, enrollment will be interrupted. A Safety Monitoring Committee (SMC) will review safety data (including demographics, adverse events, serious adverse events, adverse events of special interest, and relevant laboratory data). The SMC will then provide a recommendation as to whether the study may continue, whether amendment(s) to the protocol should be implemented, or whether the study should be stopped. Recruitment will only be resumed accordingly to SMC decision.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient/legal representative before performing any protocol-related procedures, including screening evaluations.
* Patient state to comply with all the study procedures and treatments. Patients must be accessible for treatment and follow-up. Patients registered for this trial must be treated and followed at the participating Centre.
* Age ≥ 18 years at the time of informed consent.
* ECOG Performance Status ≤ 2.
* Life expectancy of ≥ 3 months.
* Have histologically documented adenocarcinoma of the colon or rectum, which is initially metastatic or unresectable locally advanced.
* Subjects must be willing to provide the most recently available formalin-fixed paraffin-embedded tumor tissue blocks (or at least 25 freshly sectioned slides) for translational analyses (sampled before 1st treatment course). If archival tissue is not available for HER2 testing or for exploratory aims, then a newly obtained baseline biopsy of an accessible tumor lesion is required before Cycle 1 Day 1 timeframe. Biopsy must contain adequate tissue for analysis; the following biopsy types are acceptable: resection, excision, punch (skin lesions only) and core needle biopsies.
* Presence of locally determined HER2 overexpression/amplification defined as IHC 3+ or 2+/ISH amplified on archival/newly obtained tumor tissue, according to the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines for gastric/gastroesophageal cancer.
* Have RAS known status and pMMR/MSS status by standard local testing.
* Have radiographically measurable disease per RECIST v1.1.
* Have adequate hematological, hepatic, renal, cardiac and coagulation function, as defined below, obtained ≤ 7 days prior to enrollment (Cycle 1 Day 1):

  * Absolute neutrophil count (ANC) ≥ 1500/mm3. (Granulocyte-colony stimulating factor administration is not allowed within 1 week prior to C1D1).
  * Platelet count ≥ 100000/mm3. (Platelet transfusion is not allowed within 1 week prior to C1D1)
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN (≤ 5 x ULN if liver metastases are present).
  * Serum albumin ≥ 2.5 g/dL.
  * Creatinine clearance ≥ 60 mL/min as determined by Cockcroft-Gault (using actual body weight).
  * Left ventricular ejection fraction (LVEF) ≥ 50% within 28 days before enrollment.
  * International normalized ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 x ULN.
* Have had adequate washout period from previous treatment before screening, defined as:

  * ≥ 4 weeks from major surgery.
  * ≥ 4 weeks from radiation therapy, including palliative stereotactic radiation therapy to the chest.
  * ≥ 3 weeks from anti-cancer chemotherapy [immunotherapy (non-antibody-based therapy)], retinoid therapy, hormonal therapy.
  * ≥ 4 weeks from antibody-based anti-cancer therapy
  * ≥ 2 weeks or 5 half-lives (whichever is longer) from targeted agent- and small molecule-based therapy
  * ≥ 6 weeks from nitrosureas or mitomycin C
  * ≥ 1 week from TKIs approved for treatment of patients with non-small-cell lung cancer (baseline CT must be completed after discontinuation of TKI)
  * > 2 weeks from chloroquine/hydroxychloroquine
  * ≥ 2 weeks from cell-free and Concentrated Ascites Reinfusion Therapy (CART), peritoneal shunt or drainage of ascites, pleural or pericardial effusion.
* Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta- human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of IP. Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
* Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in Table 1. From the time of screening and must agree to continue using such precautions for 7 months after the last dose of investigational product (IP). Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic, or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
* Female participants must not donate, or retrieve for their own use, ova from the time of enrolment and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.
* Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IP for T-DXd while 6 months for capecitabine and bevacizumab. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period, by employing protocol-recommended methods. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of randomization/enrollment, throughout the study and for 4 months after the last dose of IP for T-DXd while 6 months for capecitabine and bevacizumab. Preservation of sperm should be considered prior to enrollment in this study.

Exclusion Criteria:

* Have previously received any systemic anticancer therapy for CRC in the metastatic/locally advanced unresectable setting or have participated in any interventional clinical trial for CRC in the metastatic/locally advanced unresectable setting. Subjects may have received prior fluoropyrimidine with or without oxaliplatin for CRC in the adjuvant or neoadjuvant setting if it was completed > 6 months before enrollment.
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment.
* Have previously been treated with an anti-HER2 agent and/or a topoisomerase I inhibitor.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medications.
* Have substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
* Patients with a medical history of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV). Subjects with troponin levels above ULN at screening (as defined by the manufacturer) and without any myocardial-related symptoms should undergo a cardiologic consultation before enrollment to rule out MI.
* Corrected QT interval (QTcF) prolongation to > 470 msec (females) or > 450 msec (males) based on average of the screening 12-lead ECG.
* Symptomatic arterial hypertension or uncontrolled arterial hypertension, as determined by the investigator.
* Have a history of (non-infectious) ILD/pneumonitis that required steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g., severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc.).
* Any autoimmune, connective tissue, or inflammatory disorders (e.g., Rheumatoid arthritis, Sjögren's, sarcoidosis etc.) where there is documented, or a suspicion of, pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
* Prior pneumonectomy (complete).
* A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).
* Have unresolved toxicities from previous anticancer therapy, defined as toxicity (other than alopecia) not yet resolved to Grade ≤ 1 or baseline. Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to Grade > 2 for at least 3 months before enrollment/cycle 1 day 1 and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy such as: chemotherapy-induced neuropathy and fatigue.
* Patients with known hypersensitivity to the study drug or to its excipients.
* Patients with known hypersensitivity to other monoclonal antibodies.
* Pregnant or breastfeeding female patients, or patients who are planning to become pregnant. Sexually active men not willing to use adequate contraception during whole study period.
* Previous or concurrent malignancy within 3 years of study entry. Exceptions are adequately resected non-melanoma skin cancer, curatively treated in-situ diseases, and other solid tumors that have been curatively treated.
* Presence of any of the following dihydropyrimidine dehydrogenase (DPYD) polymorphism, based on local laboratory testing: DPYD 2a (c.1905+1G>A); DPYD13 (c.1679 T>G); DPYD D949V (c.2846 A>T). French and German patients may undergo baseline uracilemia assessment as detailed below in spite of polymorphism testing.
* Have a history of transient ischemic attack, cerebrovascular accident, myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or cardiac surgery within 6 months prior to enrollment (Cycle 1 Day 1).
* Have a history of a significant bleeding event (e.g., bleeding needing medical intervention) within 6 months prior to enrollment (Cycle 1 Day 1) unless the source of bleeding has been definitively treated.
* Have a history of GI perforation within 12 months prior to enrollment (Cycle 1 Day 1).
* Major surgical procedure or significant traumatic injury ≤ 28 days prior to enrollment (≤ 56 days for hepatectomy, open thoracotomy or major neurosurgery) or anticipation of need for major surgical procedure during the course of the study.
* Serious, non-healing wound, ulcer, or bone fracture.
* Prior organ transplantation, including allogenic stem-cell transplantation.
* Known history of HIV infection.
* Active infection including tuberculosis, hepatitis B, hepatitis C. Patients positive for hepatitis C (HCV) antibody are eligible only if HCV RNA polymerase chain reaction (PCR) is negative. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible only if meeting the following criteria:

  * HBsAg negativity (for more than 6 months off anti-viral treatment).
  * Anti-HBc positivity (IgG or total Ig).
  * Absence of cirrhosis or fibrosis on prior imaging or biopsy.
  * Absence of HCV co-infection and no history of HCV co-infection.
  * Access to a local HBV expert during and after the study Patients meeting all abovementioned criteria must be closely monitored for HBV reactivation.
* Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent and that would limit compliance with trial requirements.
* Use of any disallowed drugs (see Section 7.5).

Additional exclusion criteria for France and Germany:

* Patients with dihydropyrimidine dehydrogenase (DPD) enzyme deficiency (uracilemia ≥ 16 ng/mL)
* Patient who is under judicial protection and patient who is legally institutionalized or under guardianship or not able to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 24 months
  Overall response rate will be defined as the proportion of patients who achieve either a partial or complete response as best responses to study treatment according to RECIST v1.1 criteria. Response will be assessed as per blinded independent central review

SECONDARY OUTCOMES:
Progression-free survival | 24 months
  Progression-free survival is defined as the time from treatment start to radiological evidence of disease progression (as per RECIST v1.1 criteria) or death, whichever occurs first. PFS will be assessed by BICR and Investigator-assessed.
Overall survival | 48 months
  Overall survival is defined as the time from treatment start to death.
Treatment safety | 24 months
  Treatment safety is defined as the incidence of adverse events during treatment and follow-up, assessed according to CTCAE v5.0.
Disease control rate | 24 months
  Disease control rate (DCR) by BICR and Investigator assessment, defined as the proportion of subjects achieving a complete response (CR), partial response (PR) or stable disease (SD) as best response during study treatment, as per RECIST v1.1.
Early tumor shrinkage | 24 months
  Early tumor shrinkage (ETS), defined as the proportion of patients achieving a reduction in tumor size of at least 20% at first radiological reassessment.
Duration of response | 24 months
  Duration of response (DOR), defined as the time from first radiological evidence of complete or partial response to disease progression or death whichever occurs first.
Depth of response | 24 months
  Depth of response (DoR) defined as the maximum percentage of tumor shrinkage at best response relative to baseline.
CEA dynamics | 24 months
  Serum carcinoembryonic antigen (CEA) concentration will be measured in peripheral blood using standard-of-care clinical laboratory immunoassays performed at participating sites. The unit of measure will be ng/mL. CEA kinetics will be summarized as: (i) absolute CEA values (ng/mL) over time; (ii) change from baseline (absolute and percent change); and (iii) CEA normalization (conversion to within institutional normal range) when applicable. CEA dynamics will be assessed at baseline, every 9 (+/-1) weeks during treatment, at EOT and during follow-up visits through 24 months. Associations will be explored between CEA kinetics and efficacy/activity outcomes including objective response (per RECIST v1.1), duration of response, progression-free survival and overall survival, using correlation/association analyses
Central review of HER-2 status | 24 month
  Tumor HER2 status will be centrally assessed on archival tumor tissue on which local HER-2 positivity was assessed. HER-2 testing will be performed by means of immunohistochemistry (IHC) assay with in situ hybridization (ISH) in case of IHC 2+ scores. HER2 status will be evaluated according to the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines for gastric/gastroesophageal cancer. The measure will be reported as HER2 IHC score category, ISH result (where applicable), and overall central HER2 status (positive vs negative). Concordance between central and local HER2 results will be evaluated using percent agreement (overall/positive/negative agreement as applicable) and Cohen's kappa statistic. Exploratory associations between centrally confirmed HER2 status (and/or HER2 categories) and efficacy/activity outcomes (objective response per RECIST v1.1, progression-free survival, overall survival) will be assessed.
Quality of life as assessed by the European Organization for Research and Treattment of Cancer (EORTC) QLQ-C30 | 24 months
  Quality of life will be assessed through Patients reported outcomes (completion of quality-of-life questionnaires, European Organization for Research and Treattment of Cancer (EORTC) QLQ-C30 during treatment). Questionnaires will be administered at baseline, every 9 weeks +/- 7 days during treatment and at the end of treatment.
CA19.9 dynamics | 24 months
  Serum carbohydrate antigen 19-9 (CA19-9) concentration will be measured in peripheral blood using standard-of-care clinical laboratory immunoassays performed at participating sites. The unit of measure will be U/mL. CA19-9 kinetics will be summarized as: (i) absolute CA19-9 values (U/mL) over time; (ii) change from baseline (absolute and percent change); and (iii) CA19-9 normalization (conversion to within institutional normal range) when applicable. CA19-9 dynamics will be assessed at baseline, every 9 (+/- 1) weeks during treatment, at EOT and during follow-up visits through 24 months. Associations will be explored between CA19-9 kinetics and efficacy/activity outcomes including objective response (per RECIST v1.1), duration of response, progression-free survival and overall survival, using correlation/association analyses.
Quality of life as assessed by the European Organization for Research and Treattment of Cancer (EORTC) QLQ-CR-29 | 24 months
  Quality of life will be assessed through Patients reported outcomes (completion of quality-of-life questionnaires, European Organization for Research and Treattment of Cancer (EORTC) QLQ-CR-29 during treatment). Questionnaires will be administered at baseline, every 9 weeks +/- 7 days during treatment and at the end of treatment.
Quality of life as assessed by the European Organization for Research and Treattment of Cancer (EORTC) EuroQol EQ-5D | 24 months
  Quality of life will be assessed through Patients reported outcomes (completion of quality-of-life questionnaires, European Organization for Research and Treattment of Cancer (EORTC) EuroQol EQ-5D during treatment). Questionnaires will be administered at baseline, every 9 weeks +/- 7 days during treatment and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (28):
- France (5):
  - Hopital Prive Jean Mermoz, Lyon
  - Hôpital La Timone - APHM, Marseille
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universitaire Reims, Reims
  - Groupe Hospitalier Rance Emeraude, St-Malo
- Germany (2):
  - Charite Universitaetsmedizin, Berlin
  - Krankenhaus Nordwest, Frankfurt
- Italy (16):
  - Istituto Tumori Bari Giovanni Paolo II, Bari, Bari
  - A.O.U Careggi, Florence, Firenze
  - Istituto Europeo Di Oncologia S.r.l., Milan, Italy
  - Azienda Unita Sanitaria Locale Della Romagna, Ravenna, Italy
  - Humanitas Mirasole S.p.A., Rozzano, Italy
  - Azienda Ospedaliera Card. G. Panico, Tricase, LE
  - Fondazione IRCCS Istituto Nazionale dei Tumori - Milano, Milan, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena, Missouri
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Policlinico Tor Vergata Roma, Roma, Roma
  - IFO-Regina Elena Institute for Cancer Research, Roma, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Udine
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Naples
  - IRCCS Istituto Nazionale Tumori "Fondazione Giovanni Pascale", Napoli
  - Fondazione IRCCS Istituto Oncologico Veneto, Padua
  - U.O. Oncologia Medica 2 Universitaria - Azienda Ospedaliero-Universitaria Pisana Dipartimento di Ricerca Traslazionale e Nuove Tecnologie - University of Pisa, Pisa
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Fundación Jiménez, Madrid
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
The trial results concerning the primary, secondary and exploratory outcomes will be published according to the standard guidelines. IPD could eventually be requested to the Sponsor and Principal Investigator, who will carefully evaluate the formal and motivated request